CLINICAL TRIAL: NCT01527955
Title: Troubleshooting the Mind Through Kelee® Meditation: A Distinctive and Effective Therapeutic Intervention for Stress, Anxiety, and Depression
Brief Title: Kelee® Meditation: A Distinctive and Effective Therapeutic Intervention for Stress, Anxiety, and Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Daniel Lee, MD, Associate Clinical Professor of Medicine, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB Project#081197
Record Dates: First submitted 2012-02-02; First posted 2012-02-07 (Estimated); Last update posted 2012-02-07 (Estimated); Status verified 2012-02

CONDITIONS: Stress; Anxiety; Depression
Keywords: Kelee; Meditation; Stress; Anxiety; Depression; Brain; Mind
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Kelee Meditation — The participants were instructed on how to perform Kelee Meditation (KM) at the initial session. This was followed by a comprehensive review of the Kelee principles and reference points over the subsequent 12 weeks. At the beginning of each weekly session, a group meditation was performed, which was followed by individual introspection and contemplation. Participants recorded their observations and experiences in a KM journal. Each participant had the opportunity to share his own journal entry and to ask questions about his own observations and experiences since starting KM. Participants were encouraged to perform the KM practice 10 minutes twice daily throughout the 12 weeks of the study.

SUMMARY:
The purpose of this study is to determine how effective Kelee meditation is in improving stress, anxiety, and depression.

DETAILED DESCRIPTION:
The Kelee and Kelee meditation (KM) were developed and founded by Ron W. Rathbun. KM is a unique and distinctive form of meditation that is easy to learn and requires only about 10 minutes twice a day to perform. The goal and discipline of KM is the development of one-pointed stillness of mind. To better comprehend how KM is effective in reducing stress, anxiety, and depression, one must understand the difference between concentration and meditation, and the basic principles of the Kelee. Experiencing and understanding the distinction between brain function and mind function are of vital importance in KM. Brain function is associated with the tension-based, intellectual, thinking process and the five physical senses whereas mind function is associated with the relaxation-based, experiential, mental feeling process, self-awareness, and clear perception. Performing KM leads to the calming of brain function and opening to the experience of mind function. With continued practice, persistence, and patience, the practitioner can begin to learn on his own how to examine and understand (ie, troubleshoot) his own thoughts and feelings from a calm, clear internal space that is free from the negative chatter and preconception associated with the brain. This increases self-awareness of the presence of internalized compartments (misperceptions of life that exist as negative thoughts and/or feelings) and the practitioner begins to develop clarity of perception. Clear perception allows one to begin the process of detachment from internalized compartments, which occurs through the cessation of looping followed by the processing of compartments. As each negative compartment dissipates, the practitioner experiences a subtle, but cumulative, corresponding improvement in stress, anxiety, and depression. When the flow of the Kelee is allowed to be, there is balance between the thinking and the feeling process leading to overall well-being, which leads to improved self-efficacy and reinforces the repetition of KM.

ELIGIBILITY:
Inclusion Criteria:

* Documented HIV-1 infection
* Ages 18 to 65
* Experiencing some level of stress, anxiety, or depression
* No current use of other meditation practices or holistic modalities

Exclusion Criteria:

* Non-English readers or speakers
* Hearing-impaired
* Low literacy below 5th grade reading and comprehension level

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2008-09; Primary Completion 2010-09 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Change in Total Score of Depression, Anxiety, and Stress Scales-42 (DASS-42) | From Week 0 (baseline) to Week 12
  The DASS is a set of 3 self-report scales designed to measure the negative emotional states of depression, anxiety and stress and to further the process of defining, understanding, and measuring the ubiquitous and clinically significant emotional states usually described as depression, anxiety and stress. Each of the 3 DASS scales contains 14 items. Subjects are asked to use 4-point severity/frequency scales to rate the extent to which they have experienced each state over the past week. Scores for Depression, Anxiety and Stress are calculated by summing the scores for the relevant items.

SECONDARY OUTCOMES:
Change in Depression Subscale Score of DASS-42 | From Week 0 (baseline) to Week 12
  The Depression scale assesses dysphoria, hopelessness, devaluation of life, self-deprecation, lack of interest/involvement, anhedonia, and inertia.
Change in Anxiety Subscale Score of DASS-42 | From Week 0 (baseline) to Week 12
  The Anxiety scale assesses autonomic arousal, skeletal muscle effects, situational anxiety, and subjective experience of anxious affect.
Change in Stress Subscale Score of DASS-42 | From Week 0 (baseline) to Week 12
  The Stress scale is sensitive to levels of chronic non-specific arousal. It assesses difficulty relaxing, nervous arousal, and being easily upset/agitated, irritable/over-reactive and impatient.
Change in Total Score of Beck Depression Inventory-II (BDI-II) | From Week 0 (baseline) to Week 12
  The BDI-II contains 21 questions, each answer being scored on a scale value of 0 to 3. The cutoffs are as follows: 0-13: minimal depression; 14-19: mild depression; 20-28: moderate depression; and 29-63: severe depression. Higher total scores indicate more severe depressive symptoms.
Change in Total Score of Beck Anxiety Inventory (BAI) | From Week 0 (baseline) to Week 12
  The BAI consists of 21 questions about how the subject has been feeling in the last week, expressed as common symptoms of anxiety. Each answer is scored on a scale value of 0 to 3. The cutoffs are as follows: 0-7: minimal anxiety; 8-15: mild anxiety; 16-25: moderate anxiety; and 26-63: severe anxiety.
Change in Total Score of Perceived Stress Scale-10 (PSS-10) | From Week 0 (baseline) to Week 12
  The Perceived Stress Scale (PSS) is a measure of the degree to which situations in one's life are appraised as stressful. Items were designed to tap how unpredictable, uncontrollable, and overloaded respondents find their lives. The scale also includes a number of direct queries about current levels of experienced stress. PSS scores are obtained by reversing responses (e.g., 0 = 4, 1 = 3, 2 = 2, 3 = 1 & 4 = 0) to the four positively stated items (items 4, 5, 7, & 8) and then summing across all scale items. Higher total scores suggest a higher degree of perceived stress.
Change in Global Severity Index (GSI) of the Symptom Checklist-90-Revised (SCL-90-R) | From Week 0 (baseline) to Week 12
  The Symptom Checklist-90-R (SCL-90-R) instrument helps to evaluate a broad range of psychological problems and symptoms of psychopathology. The instrument is also useful in measuring patient progress or treatment outcomes. The Global Severity Index (GSI) is the summary of the test and is designed to measure overall psychological distress.
Change in Mental Component Summary (MCS) of the Short Form-36 Health Survey (SF-36) | From Week 0 (baseline) to Week 12
  The SF-36 is a short-form health survey with only 36 questions. It yields an 8-scale profile of functional health and well-being scores as well as psychometrically-based physical and mental health summary measures [Physical Component Summary (PCS) and Mental Component Summary (MCS)] and a preference-based health utility index.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Lee, MD, Principal Investigator — University of California, San Diego
Locations (2):
- United States (2):
  - Being Alive San Diego, San Diego, California
  - University of California, San Diego Medical Center, San Diego, California

REFERENCES:
- See also: Kelee Foundation website for more information about Kelee Meditation — http://www.thekelee.org